CLINICAL TRIAL: NCT05706532
Title: Cardiovascular and Cerebrovascular Control in Healthy Adult Subjects
Brief Title: Cardiovascular and Cerebrovascular Control in Healthy Subjects
Acronym: CardioSan
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Vlasta Bari, Assistant Professor, PhD, IRCCS Policlinico S. Donato
Other Study IDs: CardioSan
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Autonomic Nervous System; Cerebral Autoregulation
Keywords: autonomic nervous system; heart rate variability; cerebral autoregulation; peripheral resistances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy: 60 healthy subjects; age >18; sinus rhythm; absence of autonomic diseases or dysfunctions.
  Interventions: Diagnostic Test: active standing

INTERVENTIONS:
Diagnostic Test: active standing — Data are acquired with patients resting in supine position for 10 minutes and for 10 minutes during active standing

SUMMARY:
The aim of the study is to evaluate autonomic function and cerebrovascular control in 60 healthy subjects by means of noninvasive analysis of time series variability.

To this extent, heart period, systolic and mean arterial blood pressure, cerebral blood velocity, peripheral resistances, respiration will be recorded from subjects during an orthostatic challenge.

The interactions between autonomic cardiovascular function, cerebrovascular and peripheral control will be evaluated exploiting the most advanced signal processing techniques.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* sinus rhythm
* informed consent signed

Exclusion Criteria:

* age <18
* presence of autonomic nervous system diseases or dysfunctions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the state and interactions of autonomic function and cerebrovascular control | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No